CLINICAL TRIAL: NCT02965937
Title: Effectiveness of Story-Centred Care Intervention Program in Older Persons Living in Long-term Care Facilities：A Randomised Clinical Study
Brief Title: Effectiveness of Story-Centred Care Intervention Program in Older Persons Living in Long-term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Fung-Wei Chang, Director, Head of Obstetrics and Gynecology, Clinical Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1-101-05-090
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: Attentively embracing story; story-centred care; heart rate variability; cognitive function
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Story-Centred Care Intervention Program (Experimental): A theory-guided approach that emphasises a health-promoting potential of nurse-person dialogue about a health challenge.Participants randomised to the IG will be made to participate in a 4-week long story-centred care intervention program conducted by a trained researcher.
  Interventions: Other: Story-centred care intervention program
- Health consultation control condition (Active Comparator): Participants randomised to the control group will receive a health consultation from a trained researcher once a week for 4 weeks. The health consultation will be tailored to the participants' needs. Based on a previous study, the health consultation will include pain management, healthy nutrition, how to make best use of medical services and education and counselling for individual health-related concerns.
  Interventions: Other: Health consultation control condition

INTERVENTIONS:
Other: Story-centred care intervention program — Participants in the intervention group received the "Story-Centred Care Intervention Program" once a week for four weeks.
  Arms: Story-Centred Care Intervention Program
Other: Health consultation control condition — The control group received a health consultation from researchers once a week for four weeks.. The health consultation will be tailored to the participants' needs. Based on a previous study12, the health consultation will include pain management, healthy nutrition, how to make best use of medical services and education and counselling for individual health-related concerns.
  Arms: Health consultation control condition

SUMMARY:
The study aim is to evaluate the effectiveness of Story-Centred Care Intervention Program on reducing depressive symptoms, improving cognitive function, HRV, Blood pressure and quality of life in older adults living in a long-term care facility.

DETAILED DESCRIPTION:
Design A single-blind two-group longitudinal experimental study will be conducted to compare a story-centred care intervention program with a health consultation control condition. After receiving informed consents, participants will be randomly assigned to one of the two treatment conditions, either a story-centred care intervention program or a health consultation control condition. Each intervention will be conducted for 4 weeks. Measurements will be obtained at the following time points: pre-intervention (baseline), post-intervention and 1-month- and 3-month follow-up (see Figure 1). Outcome measurements include the following parameters: 15-item geriatric depression scale test (GDS-15), short portable mental status questionnaire (SPMSQ) , WHO Quality of Life-BREF (WHOQOL-BREF), blood pressure and 5-minute HRV.

Recruitment Participants will be recruited from January 2013 to August 2013 via posters and notifications during routine activities and gatherings. The study design and protocols will be reviewed and approved by the institutional review board of the participating hospital. At the content session, all assessments and procedures will be fully explained. When participants express their interest in participating in the study, they need to leave their contact information at the front desk. The research team will contact the participants as soon as a list is compiled.

Assessment of eligibility and randomisation Participants will beconsidered eligible if they meet the inclusion criteria. All participants will be informed that they can withdraw themselves from the study at any time. Before randomisation, participants will be asked to answer a few questionnaires and will be subjected to the 5-minute HRV test. The questionnaires include demographic characteristics, the 15-item geriatric depression scale test (GDS-15) and SPMSQ. Randomisation will be conducted using a computer-generated randomisation scheme (SPSS software Version 21.0). Participants will be randomly assigned to the story-centred care intervention program or to the health consultation control condition. The random allocation sequence will be set in a uniform 1:1 allocation ratio.

Blinding Participants will be randomly assigned to either the story-centred care intervention program or the health consultation control condition. They will be informed not to disclose their randomisation status to anyone. The outcome evaluator will be blinded to the assigned condition of the participants.

Intervention Participants will randomly be assigned to the experimental (intervention) group (IG) or the control group (CG) using SPSS software (Version 21.0). Participants in the IG will receive the story-centred care intervention program once a week for 4 weeks; the CG will receive health consultation from researchers once a week for 4 weeks.

Story-centred care intervention program Participants randomised to the IG will be made to participate in a 4-week long story-centred care intervention program conducted by a trained researcher. A trained researcher will facilitate the six-step intervention. Step 1 involves gathering stories about complicated health challenges of the participants. the investigators will guide the participants in describing their health challenges using elements of a story. The challenges include current health problems, past experiences related to these problems and expectations for dealing with these problems. During Step 2, connections of the health challenges to existing literature will be made and a story is reconstructed. In order to ensure that the health challenge is a true reflection of participants' condition, the investigators identifies the complicated health challenges of the participants through existing literature and helps them revise the story to identify their most important and influential health challenges. Step 3 determines key moments of the health challenges by understanding the participants' feelings about these challenges. Step 4 involves accepting the story episodes, which will be recorded and consolidated into a theme for the entire story. In Step 5, the researcher guides the participant to describe approaches that can motivate him/her to resolve existing health challenges. In Step 6, the participant is encouraged to resolve the challenges by generating new meanings of life to improve their overall well-being. During the process, the researcher does not interfere but asks questions to help the participants clarify vague parts of the health story.

Health consultation control condition Participants randomised to the control group will receive a health consultation from a trained researcher once a week for 4 weeks. The health consultation will be tailored to the participants' needs. Based on a previous study, the health consultation will include pain management, healthy nutrition, how to make best use of medical services and education and counselling for individual health-related concerns.

Statistical analysis The investigators will use descriptive statistics (mean, standard deviation, frequency and percentage) to analyse participant characteristics and primary outcomes. Mann-Whitney U test is used to examine the continuous variables between groups and chi-square test (or Fisher's Exact tests where appropriate) is used to examine the categorical variables between groups. Generalised estimating equation (GEE) is used to examine the effects of the story-centred care intervention program on the improvement of depression, cognitive function, quality of life, blood pressure and HRV. The SPSS 21.0 software package, Chinese version, will be used to analyse the data. All tests are two-tailed and α < 0.05 is considered statistically significant.

Sample size calculation Sample size will be estimated using a repeated-measures MANOVA approach, within-between interaction in G*power 3.0.10 with power = 0.8, type 1 error α = 0.05 and effect size η2 = 0.43. We will require a sample size of 64 (32 per group) rising to 70 accounting for a 10% loss in follow-up.

Outcomes measurements

Primary outcome 15-item geriatric depression scale test (GDS-15): The GDS-15 test assesses depressive symptoms. The GDS-15 test is a self-administered questionnaire with a yes/no response. This study used the Chinese version of the GDS-15 test. A higher score indicates more severe depression with a sensitivity of 70.6% and a specificity of 70.1% for older adults.

Secondary outcome The short portable mental status questionnaire (SPMSQ): The SPMSQ assesses disorientation, personal profile, short- and long-term memory and computing ability. The number of incorrect answers indicates the level of cognitive function. This study uses the Chinese version of the SPMSQ. To suit the context of this study, some items are deleted, resulting in a 10-item questionnaire scored as follows: 0-2, intact cognitive function; 3-4, mild cognitive impairment and ≥5, moderate to severe cognitive impairment. The test-retest reliability of the Chinese SPMSQ for older adults is 0.714.

Heart rate variability (HRV): HRV is measured using the CheckMyHeart handheld HRV device (DailyCare BioMedical Inc., Chungli, Taiwan), which is a limb-lead ECG (modified lead I) recorder with HRV analytical software. It is CE certified in several countries (US, Canada, Japan and Taiwan) and has been used in previous studies. The investigators make use of HRV time-domain parameters of standard deviation of the normal-to-normal intervals (SDNN) and root mean square of successive differences (RMSSD) as outcome variables, which are more strongly associated with psychological measures than frequency domain.

WHO Quality of Life-BREF(WHOQOL-BREF):The WHOQOL-BREF includes 26 questions covering four domains: physical health, psychological health, social relationships, and environment. Two items have been added to the Taiwanese version in order to reflect Taiwanese cultural differences, bringing the total number of items to 28. The two questions are 'Do participants feel respected by others?' and 'Are participants usually able to get the food (i.e. lack of availability) that participants like?' Each item is scored from 1 to 5, and the higher the score, the greater the perceived quality of life. Scores are transformed linearly into a 28-140 possible range so that a mean scale score can be calculated. Cronbach's alpha is above 0·69 for all subscales (range 0·69-0·87) and 0·93 for the whole scale in the present study.

ELIGIBILITY:
* Inclusion Criteria:
* - those who are ≥65 years old and live in long-term care facilities
* - have clear consciousness and normal hearing and conversation capability
* - are not taking any antidepressants at the time of the study
* - are not clinically diagnosed with dementia or have an SPMSQ score of ≥5
* - have not lost a loved one in the past 3 months and
* Exclusion Criteria:
* -meet DSM-IV criteria for Dementia of the Alzheimer's type
* -suffer from moderate to severe cognitive impairment (SPMSQ > 5)
* -are taking antidepressants at the time of the study
* -are undergoing other psychotherapy during the study and
* -have any underlying medical illness that could interfere with the treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
15-Item Geriatric Depression Scale | Change from depressive symptoms at 4 months

SECONDARY OUTCOMES:
The Short Portable Mental Status Questionnaire | Change from cognitive at 4 months
blood pressure | Change from blood pressure at 4 months
Heart rate variability | Change from HRV at 4 months
WHO quality of life-BREF | Change from quality of life at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kao Chi-Wen, PHD, Study Director — Taiwan Nurses Association

IPD SHARING:
Plan to Share IPD: No